CLINICAL TRIAL: NCT05840458
Title: Effect of Systemic Analgesia and Systemic Analgesia Associated With Pericapsular Nerve Block in Proximal Femoral Fractures
Brief Title: Pericapsular Nerve Block in Proximal Femoral Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Sponsor
Other Study IDs: 48721715.0.0000.5461
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-04

CONDITIONS: Femoral Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PENG Block: Patients will be submitted to PENG block intervention guiding by ultrasound.
  Interventions: Procedure: PENG Block

INTERVENTIONS:
Procedure: PENG Block — Patient will be placed in the supine position and the ultrasound probe will be placed in the transverse plane over the anterior inferior iliac spine (AIIS) and aligned with the pubic ramus by rotating the probe counterclockwise by approximately 45 degrees. A 22-gauge, 100 mm needle will be inserted using the plane approach from lateral to medial, between the psoas tendon anteriorly and the pubic ramus posteriorly. Following a negative aspiration, 20 mL of 0.375% ropivacaine will be injected. The needle position will be confirmed by visualizing the separation of layers with the dispersion of the injected volume.

SUMMARY:
Proximal femoral fractures commonly occur above 50 years and regional anesthesia could be a complement in the perioperative treatment of the patients. The use of pericapsular nerve group block (PENG Block) has been proposed to reduce pain. However, no studies have explored the efficient of the systemic analgesia associated with PENG Block in functional limitation in the preoperative period. In this sense, the main goal of this study is to evaluate the effectiveness of systemic analgesia associated with PENG Block in patients with proximal femoral fractures in the period preceding the surgical procedure.

DETAILED DESCRIPTION:
Focus on functional capacity will be measured by the Activity Measure for Post-Acute Care (AM-PAC) short version of the "6 Clicks", pain intensity will be assessed using the numerical rating scale, and opioid consumption. This study will include 21 patients admitted to the Emergency Room with proximal femoral fractures.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral proximal femoral fractures admitted to the emergency room of the Hospital Sírio-Libanes,
* aged 18-105 years
* with the American Society of Anesthesiology (ASA) physical status I, II, or III.

Exclusion Criteria:

* allergy to metamizole and/or ropivacaine
* history of mental disorders
* presence of chronic pain as assessed using the Douleur Neuropathique 4 (DN4) questionnaire

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral proximal femoral fractures admitted to the emergency room.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional impairment | Before the intervention
  The Short-form of Activity Measure for Post-Acute Care (AM-PAC- "6 clicks") is a measure of basic patient mobility will be used. Higher scores mean better outcomes. Minimum 6 points, maximum 26 points.
Functional impairment | 12 hours after intervention
  The Short-form of Activity Measure for Post-Acute Care (AM-PAC- "6 clicks") is a measure of basic patient mobility will be used. Higher scores mean better outcomes. Minimum 6 points, maximum 26 points.

SECONDARY OUTCOMES:
Pain levels | Before performing the PENG block
  The Numeric Rating Scale will be used to evaluate pain levels. Higher scores mean worst. outcomes. Minimum 0 point, maximum 10 points.
Pain levels | 1 hour after performing the PENG block
  The Numeric Rating Scale will be used to evaluate pain levels. Higher scores mean worst. outcomes. Minimum 0 point, maximum 10 points.
Pain levels | 12 hours after performing the PENG block
  The Numeric Rating Scale will be used to evaluate pain levels. Higher scores mean worst. outcomes. Minimum 0 point, maximum 10 points.
Opioid consumption | 24 hours after performing the PENG Block
  The total opioid consumption will be evaluated 24 hours after performing the PENG Block

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio-Libanês, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Membership of the Working Party; Griffiths R, Alper J, Beckingsale A, Goldhill D, Heyburn G, Holloway J, Leaper E, Parker M, Ridgway S, White S, Wiese M, Wilson I. Management of proximal femoral fractures 2011: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2012 Jan;67(1):85-98. doi: 10.1111/j.1365-2044.2011.06957.x. PMID 22150501
- [Background] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- [Background] Hua H, Xu Y, Jiang M, Dai X. Evaluation of Pericapsular Nerve Group (PENG) Block for Analgesic Effect in Elderly Patients with Femoral Neck Fracture Undergoing Hip Arthroplasty. J Healthc Eng. 2022 Feb 9;2022:7452716. doi: 10.1155/2022/7452716. eCollection 2022. PMID 35186238